CLINICAL TRIAL: NCT00520247
Title: Efficacy of Antihypertensive and Plasma Total Homocysteine Lowering Combined Therapy With Enalapril and Folic Acid in Hypertensive Patients:A Multicenter Double Blind Randomized Clinical Trial
Brief Title: Effect of Enalapril Plus Folic Acid on Blood Pressure and Glycometabolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Medical University (Other)
Collaborators: Peking University First Hospital (Other); Huashan Hospital (Other); Harbin Medical University (Other); China Medical University Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005L01101
Record Dates: First submitted 2007-08-17; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Plasma Total Homocysteine Level; Blood Pressure
Keywords: enalapril; folic acid; hyperglycemia; hypertension; fasting plasma glucose
MeSH Terms: conditions — Hyperglycemia; Hypertension | interventions — Enalapril; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: enalapril plus folic acid — enalapril 10.0 mg daily for 8 weeks (the control group); enalapril 10.0 mg plus folic acid 0.4 mg daily for 8 weeks (Low-dose group); enalapril 10.0 mg plus folic acid 0.8 mg daily for 8 weeks (High-dose group)

SUMMARY:
Combinded therapy with folic acid and enalapril may significantly decrease plasma total homocysteine level and had beneficial effect on blood pressure reduction and glycometabolism.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Age≥18 years and less than 75 years
2. Essential hypertension patients
3. Sedentary systolic blood pressure≥140mmHg and less than 180mmHg, and/or sedentary diastolic blood pressure≥90mmHg and less than 110mmHg
4. Reproductive women agree to take a reliable contraception measure during the trial
5. Written informed consent

Exclusion Criteria:

1. Pregnant women
2. Women within lactateion period
3. Hypersensitive to Angiotensin-Converting Enzyme Inhibitor (ACEI) or folic acid
4. Easily hypersensitiveness
5. Diagnosed secondum hypertension or skeptical secondum hypertension
6. Severe hypertension (sedentary systolic blood pressure greater than or equal to 180 mmHg and/or sedentary diastoleic blood pressure greater than or equal to 110 mmHg)
7. Severe diseases:

   * Cardiovascular system
   * Diagnosed cardia insufficiency (New York Health Association [NYHA] III level and higher)
   * Hypertrophic obstructive cardiomyopathy (HOCM)
   * Clinical significantly Valvular Disease of the Heart (VDH)
   * Acute coronary syndrome or coronary artery interventional therapy or coronary artery bypass graft within three months
   * Severe arrhythmia such as atrial flutter, atrial fibrillation, ventricular arrhythmia above Lown ?, atrioventricular block above II level, etc.
   * Alimentary system disorders
   * Active virus hepatitis
   * Any of alanine aminotransferase (ALT), aspartate aminotransferase (AST), galactosylhydroxylysyl glucosyltransferase (GGT), alkaline phosphatase (ALP), total bilirubin (TBIL), Direct Bilirubin (DB) was above 2 times of it's normal value upper limit, albumin (ALB) greater than 30 g/L
   * Stomach bulk resect and gastrojejunostomy, stomach intestine malabsorption

   Urinary system:
   * Serum creatinine greater than or equal to 200 mmol/L
   * Diagnosed stenosis of renal artery, solitary kidney
   * Renal transplantation

   Endocrine system:
   * Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (fasting glucose greater than or equal to 11.1 mmol/L)
   * Diagnosed and uncontrolled hyperthyrosis

   Respiratory system:
   * Chronic cough nervous or psyche system:
   * Transient Ischemia Attach (TIA) or stoke within 3 months
   * Severe peripheral nerve or vegetative nerve functional disturbance
   * Psyche or nervous system dysfunction
   * Drugs or alcohol dependence

   Others:
   * Malignant tumor
   * Malnutrition, haematogenesis dysfunction, etc.
8. Taking other antihypertensive drugs
9. Taking folic acid or other Vitamin B groups

Primary Outcome Measures:

1. Blood pressure of study participants was measured at baseline, 2th week, 4th week, 6th week and at the end of trial
2. Subjects' plasma total homocysteine concentration were measured at baseline, 4th week and at 8th week.

Secondary Outcome Measures:

1. Participants' living habit and life style were collected at baseline with the original questionnaires.
2. A follow up questionnaire was sent out at 2th week, 4th week, 6th week and at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years and less than 75 years
* Essential hypertension patients
* Sedentary systolic blood pressure≥140mmHg and less than 180mmHg, and/or sedentary diastolic blood pressure≥90mmHg and less than 110mmHg
* Reproductive women agree to take a reliable contraception measure during the trial
* Written informed consent

Exclusion Criteria:

* Pregnant women
* Women within lactateion period
* Hypersensitive to angiotensin-converting enzyme inhibitor (ACEI) or folic acid
* Easily hypersensitiveness
* Diagnosed secondum hypertension or skeptical secondum hypertension
* Severe hypertension (sedentary systolic blood pressure≥180mmHg and/or sedentary diastoleic blood pressure≥110mmHg)

Severe diseases:

* Cardiovascular system:

  * Diagnosed cardia insufficiency (NYHAⅢ level and higher)
  * Hypertrophic obstructive cardiomyopathy (HOCM)
  * Clinical significantly valvular disease of the heart (VDH)
  * Acute coronary syndrome or coronary artery interventional therapy or coronary artery bypass graft within three months
  * Severe arrhythmia such as atrial flutter, atrial fibrillation, ventricular arrhythmia above Lown Ⅱ, atrioventricular block above Ⅱ level, et al
* Alimentary system:

  * Active virus hepatitis
  * Any of alanine aminotransferase (ALT), aspartate aminotransferase (AST), galactosylhydroxylysyl glucosyltransferase (GGT), alkaline phosphatase (ALP), total bilirubin (TBIL), direct bilirubin (DB) was above 2 times of it's normal value upper limit, albumin (ALB)>30g/L
  * Stomach bulk resect and gastrojejunostomy, stomach intestine malabsorption
* Urinary system:

  * Serum creatinine≥200mmol/L
  * Diagnosed stenosis of renal artery, solitary kidney
  * Renal transplantation
* Endocrine system:

  * Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (fasting glucose≥11.1mmol/L)
  * Diagnosed and uncontrolled hyperthyrosis
* Respiratory system:

  * Chronic cough
  * Nervous or psyche system
  * Transient ischemia attach (TIA) or stoke within 3 months
  * Severe peripheral nerve or vegetative nerve functional disturbance
  * Psyche or nervous system dysfunction
  * Drugs or alcohol dependence
* Others:

  * Malignant tumor, malnutrition, haematogenesis dysfunction, et al
  * Taking other antihypertensive drugs
  * Taking folic acid or other Vitamin B groups

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2005-09; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Blood pressure of study participants was measured at baseline, 2th week, 4th week, 6th week and at the end of trial Subjects' plasma total homocysteine concentration were measured at baseline, 4th week and at 8th week. | 8 weeks

SECONDARY OUTCOMES:
Participants' living habit and life style were collected at baseline with the original questionnaires. A follow up questionnaire was sent out at 2th week, 4th week, 6th week and at the end of the trial. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liu, Dr., Study Director — Peking University First Hopital
Locations (1):
- Inistitute for Biomedicine, Anhui Medical University, Hefei, Anhui, China